CLINICAL TRIAL: NCT04974554
Title: Clinical Trial of the Fit Families Multicomponent Obesity Intervention for African American Adolescents and Their Caregivers: Next Step From the ORBIT Initiative
Brief Title: FIT Families Multicomponent Obesity Intervention for African American Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Florida State University (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Mohan Madisetti, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00106021; 161HL155793-01 (Other Grant/Funding Number: National Heart, Lung, and Blood Institute (NHLBI)); 4R33HL155793-02 (NIH)
Record Dates: First submitted 2021-06-22; First posted 2021-07-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Obesity, Childhood; Metabolic Syndrome
Keywords: obesity, African American adolescents
MeSH Terms: conditions — Pediatric Obesity; Metabolic Syndrome; Obesity

STUDY DESIGN:
Intervention Model Description: The proposed study follows a 2 (condition: FIT Families [FIT], and HBFS x 4 (time: baseline [T1], 3-month mid-treatment [T2], 6-month end of treatment [T3], and 12-months follow-up [T4]), with random assignment of 180 caregivers/youths to one of the two treatment conditions. Repeated measures of caregiver and youth percent overweight (primary outcome) and physical activity (secondary outcome) will be collected at baseline (T1), and each of the 3 post-randomization time points (T2-T4).
Who Masked: Participant
Masking Description: Study Biostatistician will conduct the randomization of 180 subjects, 90 subjects per condition (FIT vs. HBFS) using a 1:1 allocation ratio. Research Assistants collecting data will be kept blind to participants' randomization status to the extent possible in a behavioral clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIT Families (Experimental): 1. FIT Families is a 6 month comprehensive multicomponent family-based behavioral intervention delivered by Community Health Workers (CHWs). FIT Families integrates home-based service delivery, Motivational Interviewing (MI; intrinsic motivation), Cognitive Behavior Skills Treatment (CBST; skills acquisition), supervised physical activity (PA), and Contingency Management (CM; extrinsic motivation). Sessions occur twice weekly for the first three months, and weekly for the second three months.
  Interventions: Behavioral: FIT
- Home-Based Family Support (Active Comparator): 2. Home-based Family Support (HBFS). Adolescents and their primary caregiver randomly assigned to HBFS will receive 6 months of weekly, home-based, client-centered, non-directive supportive family counseling.
  Interventions: Behavioral: Home-Based Family Support

INTERVENTIONS:
Behavioral: FIT — FIT Families is a home-based intervention that works with youth and caregivers to lose weight and improve their health. The intervention lasts 6 months. Sessions are held twice a week for the first 3 months and then once a week for the second 3 months. These sessions will take place in home with a community health worker. In addition, participants will have the opportunity to earn prizes for completing certain intervention related tasks.
  Arms: FIT Families
Behavioral: Home-Based Family Support — Home-Based Family Support Group will receive six months of weekly family counseling in the home. The weekly visits have 3 goals: 1) provide basic education in nutrition and physical recommendations for adolescent and adult obesity; 2) assess and monitor weight, physical activity, and diet via logs; and 3) offer opportunities to discuss barriers they identify to adherence to weight loss recommendations. The HBFS CHW will also address non-weight related problems such as peer or family relationship problems during the visits.
  Arms: Home-Based Family Support

SUMMARY:
Obesity is one of the most prevalent medical problems facing children and adolescents today, particularly among African American adolescents where the rate is alarmingly high. This study will test the effectiveness of FIT Families, a multicomponent family-based behavioral intervention that is culturally tailored to meet the unique needs of African American adolescents with obesity and their caregivers, against a credible attention control condition. This study has considerable public health relevance because it is delivered by Community Health Workers, maximizing the potential for the intervention to be sustained, and may reduce obesity-related health problems for a vulnerable population of adolescents.

DETAILED DESCRIPTION:
The alarming rates of obesity among children and adults, particularly among ethnic minorities, has been identified by the National Institutes of Health as one of the most serious public health challenges facing our nation in the 21st century. South Carolina (SC), part of the "Stroke Belt," has the 3rd highest obesity rate among US children at 39.2% and the 12th highest obesity rate among US adults at 32.3%. Unfortunately, African Americans in SC are disproportionately more likely to be overweight or obese (75.7% of adults, 40% of children), which places them at considerable high-risk for obesity-related diseases such as asthma, Type 2 diabetes, cardiovascular disease, hypertension, stroke, and some forms of cancer. This public health challenge is compounded by the lack of available intervention strategies specially tailored to meet the unique needs of ethnic minorities. This R01 randomized clinical trial, informed by the results from a recently completed NHLBI/NICHD center grant ("FIT Families Project," U01HL097889; PI-Naar) that followed the National Heart, Lung, and Blood Institute, Obesity Related Behavioral Intervention Trials (ORBIT) model for developing behavioral interventions, will examine the efficacy of FIT Families compared to a credible attention control condition. Each of four evidence-based behavioral components of FIT Families (home-based services, contingency management, motivational interviewing, cognitive behavioral skills training) were culturally tailored and optimized through a proof of concept sequential multiple randomized trial that produced weight loss among African American adolescents, a large and understudied population. One hundred and eighty obese African American adolescents aged 12-17 and their primary caregiver will be randomly assigned to one of two treatment conditions: 1) FIT Families or 2) Home-Based Family Support (HBFS) attention control condition. It is predicted that FIT Families will lead to greater reductions in adolescent and caregiver percent overweight, and increases in physical activity and the use of evidence-based weight management behaviors (self-monitoring of diet and exercise). If effective, FIT Families, which was carefully developed and adapted through successive Phases of ORBIT, has the potential to reduce disparities in obesity-related diseases (cardiovascular and metabolic) by addressing multiple risk factors among African American families and their adolescent children. Thus, this project has high significance in terms of potential public health impact and reduction in obesity related healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

1. adolescents (ages 12-17) self-identifying as AA,
2. BMI≥95th percentile for age and gender
3. primary caregiver who is either overweight (BMI 25.0 to 29.9) or obese (BMI≥30) and willing to participate in treatment
4. adolescent residing primarily with the primary caregiver within 30 miles of the MUSC, and 5) adolescent and caregiver obtain PA clearance from a health care provider (see Protection of Human Subjects).

Exclusion Criteria:

1. obesity secondary to medication use for another medical condition (e.g., steroids, antipsychotics);
2. secondary to a chronic condition (e.g., Down syndrome, Prader-Willi syndrome, Cushing's syndrome).

Exclusion criteria that apply to both adolescents and caregivers are:

1. pregnancy,
2. thought disorder (e.g., schizophrenia or other psychosis), suicidal, or homicidal
3. serious cognitive impairment (e.g., inability to complete questionnaires)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Percent of body fat | Baseline
  Percent of body fat is measured using bioelectrical impedance analysis (BIA). In BIA measurement, a very weak electronic current is passed through the body by means of four electrodes placed on the dorsal surface of the hand and foot
Percent of body fat | 3-month mid-treatment
  Percent of body fat is measured using bioelectrical impedance analysis (BIA). In BIA measurement, a very weak electronic current is passed through the body by means of four electrodes placed on the dorsal surface of the hand and foot
Percent of body fat | 6-month end of treatment
  Percent of body fat is measured using bioelectrical impedance analysis (BIA). In BIA measurement, a very weak electronic current is passed through the body by means of four electrodes placed on the dorsal surface of the hand and foot
Percent of body fat | 12-month follow-up
  Percent of body fat is measured using bioelectrical impedance analysis (BIA). In BIA measurement, a very weak electronic current is passed through the body by means of four electrodes placed on the dorsal surface of the hand and foot
Height | Baseline
  Height in meters will be obtained using a portable stadiometer.
Height | 3-month mid-treatment
  Height in meters will be obtained using a portable stadiometer.
Height | 6-month end of treatment
  Height in meters will be obtained using a portable stadiometer.
Height | 12-month follow-up
  Height in meters will be obtained using a portable stadiometer.
Weight | Baseline
  Weight in kilograms will be assessed using a portable digital scale with the capacity to reliably obtain weights up to 600 pounds.
Weight | 3-month mid-treatment
  Weight in kilograms will be assessed using a portable digital scale with the capacity to reliably obtain weights up to 600 pounds.
Weight | 6-month mid-treatment
  Weight in kilograms will be assessed using a portable digital scale with the capacity to reliably obtain weights up to 600 pounds.
Weight | 12-month follow-up
  Weight in kilograms will be assessed using a portable digital scale with the capacity to reliably obtain weights up to 600 pounds.

SECONDARY OUTCOMES:
Percent overweight | Baseline
  Percent Overweight will be calculated as the percentage BMI above the Centers for Disease Control's (CDC's) median BMI for age and gender. Body Mass Index (BMI) in kg/m2 will subsequently be calculated and converted to BMI percentile using age and gender norms from the CDC. Body Mass Index (BMI) in kg/m2 will be calculated from in home weight and height measurements. Weight in kilograms will be assessed using a portable digital scale with the capacity to reliably obtain weights up to 600 pounds. Height in meters will be obtained using a portable stadiometer.
Percent overweight | 3 month mid-treatment
  Percent Overweight will be calculated as the percentage BMI above the Centers for Disease Control's (CDC's) median BMI for age and gender. Body Mass Index (BMI) in kg/m2 will subsequently be calculated and converted to BMI percentile using age and gender norms from the CDC. Body Mass Index (BMI) in kg/m2 will be calculated from in home weight and height measurements. Weight in kilograms will be assessed using a portable digital scale with the capacity to reliably obtain weights up to 600 pounds. Height in meters will be obtained using a portable stadiometer.
Percent overweight | 6 month end of treatment
  Percent Overweight will be calculated as the percentage BMI above the Centers for Disease Control's (CDC's) median BMI for age and gender. Body Mass Index (BMI) in kg/m2 will subsequently be calculated and converted to BMI percentile using age and gender norms from the CDC. Body Mass Index (BMI) in kg/m2 will be calculated from in home weight and height measurements. Weight in kilograms will be assessed using a portable digital scale with the capacity to reliably obtain weights up to 600 pounds. Height in meters will be obtained using a portable stadiometer.
Percent overweight | 12 month follow-up
  Percent Overweight will be calculated as the percentage BMI above the Centers for Disease Control's (CDC's) median BMI for age and gender. Body Mass Index (BMI) in kg/m2 will subsequently be calculated and converted to BMI percentile using age and gender norms from the CDC. Body Mass Index (BMI) in kg/m2 will be calculated from in home weight and height measurements. Weight in kilograms will be assessed using a portable digital scale with the capacity to reliably obtain weights up to 600 pounds. Height in meters will be obtained using a portable stadiometer.
Physical activity | baseline
  Physical activity is assessed using the compact FitBit Flex2 accelerometer, which utilizes a tri-axial accelerometer and digital filtering proprietary machine-learning algorithms to analyze and estimate human movement patterns
Physical activity | 3-month mid-treatment
  Physical activity is assessed using the compact FitBit Flex2 accelerometer, which utilizes a tri-axial accelerometer and digital filtering proprietary machine-learning algorithms to analyze and estimate human movement patterns
Physical activity | 6-month end of treatment
  Physical activity is assessed using the compact FitBit Flex2 accelerometer, which utilizes a tri-axial accelerometer and digital filtering proprietary machine-learning algorithms to analyze and estimate human movement patterns
Physical activity | 12-month follow-up
  Physical activity is assessed using the compact FitBit Flex2 accelerometer, which utilizes a tri-axial accelerometer and digital filtering proprietary machine-learning algorithms to analyze and estimate human movement patterns
Self-monitoring of physical activity (PA) | Daily for six months during treatment
  Self-Monitoring of PA is assessed using daily diary logbooks completed on line
Self-monitoring of Dietary Intake | Daily for six months during treatment
  Self-Monitoring of Dietary Intake is assessed using daily diary logbooks completed on line
Symptoms of Metabolic Syndrome | Baseline
  Blood samples are obtained after a 10-12 hour fast for measurement of plasma glucose, high-density lipoprotein cholesterol (HDL-C), and triglyceride levels. Blood glucose and lipid levels are measured using the Alere Cholestech LDX, a psychometrically sound point of care analyzer that requires only one drop of whole blood.
Symptoms of Metabolic Syndrome | Baseline
  Blood pressure is measured with a sphygmomanometer 3 times, with the second and third measurement averaged for analysis.
Symptoms of Metabolic Syndrome | 3-month mid-treatment
  Blood samples are obtained after a 10-12 hour fast for measurement of plasma glucose, high-density lipoprotein cholesterol (HDL-C), and triglyceride levels. Blood glucose and lipid levels are measured using the Alere Cholestech LDX, a psychometrically sound point of care analyzer that requires only one drop of whole blood.
Symptoms of Metabolic Syndrome | 3-month mid-treatment
  Blood pressure is measured with a sphygmomanometer 3 times, with the second and third measurement averaged for analysis.
Symptoms of Metabolic Syndrome | 6-month end of treatment
  Blood samples are obtained after a 10-12 hour fast for measurement of plasma glucose, high-density lipoprotein cholesterol (HDL-C), and triglyceride levels. Blood glucose and lipid levels are measured using the Alere Cholestech LDX, a psychometrically sound point of care analyzer that requires only one drop of whole blood.
Symptoms of Metabolic Syndrome | 6-month end of treatment
  Blood pressure is measured with a sphygmomanometer 3 times, with the second and third measurement averaged for analysis.
Symptoms of Metabolic Syndrome | 12-month follow-up
  Blood samples are obtained after a 10-12 hour fast for measurement of plasma glucose, high-density lipoprotein cholesterol (HDL-C), and triglyceride levels. Blood glucose and lipid levels are measured using the Alere Cholestech LDX, a psychometrically sound point of care analyzer that requires only one drop of whole blood.
Symptoms of Metabolic Syndrome | 12-month follow-up
  Blood pressure is measured with a sphygmomanometer 3 times, with the second and third measurement averaged for analysis.
Hemoglobin A1c (HbA1c) | Baseline
  HbA1c is obtained using the Accubase A1c test kit,102 and FDA approved test that uses a capillary tube blood collection method instead of venipuncture.
Hemoglobin A1c (HbA1c) | 3-month mid-treatment
  HbA1c is obtained using the Accubase A1c test kit,102 and FDA approved test that uses a capillary tube blood collection method instead of venipuncture.
Hemoglobin A1c (HbA1c) | 6-month end of treatment
  HbA1c is obtained using the Accubase A1c test kit,102 and FDA approved test that uses a capillary tube blood collection method instead of venipuncture.
Hemoglobin A1c (HbA1c) | 12-month follow-up
  HbA1c is obtained using the Accubase A1c test kit,102 and FDA approved test that uses a capillary tube blood collection method instead of venipuncture.
Flanker task | Baseline
  Objective sub tests measuring attention and executive functioning. Scores range from 0 to 30, and the total score is used as an outcome.
Flanker task | 6-month end of treatment
  Objective sub tests measuring attention and executive functioning. Scores range from 0 to 30, and the total score is used as an outcome.
Flanker task | 12-month follow-up
  Objective sub tests measuring attention and executive functioning. Scores range from 0 to 30, and the total score is used as an outcome.
List Sorting test | Baseline
  Measures working memory. List Sorting scores are based upon a sum of the total correct across both lists which comprise the List Sorting Total Score. The raw sum score is then transformed to a standardized t-metric (mean=50, 50 and SD=10).
List Sorting test | 6-month end of treatment
  Measures working memory. List Sorting scores are based upon a sum of the total correct across both lists which comprise the List Sorting Total Score. The raw sum score is then transformed to a standardized t-metric (mean=50, 50 and SD=10).
List Sorting test | 12-month follow-up
  Measures working memory. List Sorting scores are based upon a sum of the total correct across both lists which comprise the List Sorting Total Score. The raw sum score is then transformed to a standardized t-metric (mean=50, 50 and SD=10).
Delayed Reward Discounting Task | Baseline
  Assess degree of preference for immediate over delayed rewards. The protocol is scored by by calculating where the respondent's answers place him/her amid reference discounting curves, where placement amid steeper curves indicates higher levels of impulsivity.
NEURO-QOL | 6-month end of treatment
  self-report about concerns about cognitive functioning over the previous week; quality of life. Neuro-QOL uses a T score which has a mean of 50 and the standard deviation of 10, based on the norming sample used. All Neuro-QOL banks and scales are scored such that a high score reflects more of what is being measured.
Delayed Reward Discounting Task | 6-month end of treatment
  Assess degree of preference for immediate over delayed rewards. The protocol is scored by by calculating where the respondent's answers place him/her amid reference discounting curves, where placement amid steeper curves indicates higher levels of impulsivity.
Delayed Reward Discounting Task | 12-month follow-up
  Assess degree of preference for immediate over delayed rewards. The protocol is scored by by calculating where the respondent's answers place him/her amid reference discounting curves, where placement amid steeper curves indicates higher levels of impulsivity.
NEURO-QOL | Baseline
  self-report about concerns about cognitive functioning over the previous week; quality of life. Neuro-QOL uses a T score which has a mean of 50 and the standard deviation of 10, based on the norming sample used. All Neuro-QOL banks and scales are scored such that a high score reflects more of what is being measured.
NEURO-QOL | 12-month follow-up
  self-report about concerns about cognitive functioning over the previous week; quality of life. Neuro-QOL uses a T score which has a mean of 50 and the standard deviation of 10, based on the norming sample used. All Neuro-QOL banks and scales are scored such that a high score reflects more of what is being measured.
Brief Symptom Inventory | Baseline
  Caregiver psychological symptoms. Each item of individual psychological stress is answered on a 5-point scale, ranging from 0 = not at all to 4 = extremely, with higher scores indicating more distress.
Brief Symptom Inventory | 6-month mid-treatment
  Caregiver psychological symptoms. Each item of individual psychological stress is answered on a 5-point scale, ranging from 0 = not at all to 4 = extremely, with higher scores indicating more distress.
Brief Symptom Inventory | 12-month end of treatment
  Caregiver psychological symptoms. Each item of individual psychological stress is answered on a 5-point scale, ranging from 0 = not at all to 4 = extremely, with higher scores indicating more distress.
PROMIS - Pediatric Short Form v1.0 - Depressive Symptoms | Baseline
  Adolescent depressive symptoms. The final score is represented by the T -score, that has a mean of 50 and a standard deviation of 10. With higher scores indicating more depression.
PROMIS - Pediatric Short Form v1.0 - Depressive Symptoms | 6-month mid-treatment
  Adolescent depressive symptoms. The final score is represented by the T -score, that has a mean of 50 and a standard deviation of 10. With higher scores indicating more depression.
PROMIS - Pediatric Short Form v1.0 - Depressive Symptoms | 12-month follow-up
  Adolescent depressive symptoms. The final score is represented by the T -score, that has a mean of 50 and a standard deviation of 10. With higher scores indicating more depression.
PROMIS - Pediatric Short Form v1.0 - Anxiety Symptoms | Baseline
  Adolescent anxiety symptoms. The final score is represented by the T -score, that has a mean of 50 and a standard deviation of 10. With higher scores indicating more anxiety.
PROMIS - Pediatric Short Form v1.0 - Anxiety Symptoms | 6-month end of treatment
  Adolescent anxiety symptoms. The final score is represented by the T -score, that has a mean of 50 and a standard deviation of 10. With higher scores indicating more anxiety.
PROMIS - Pediatric Short Form v1.0 - Anxiety Symptoms | 12-month follow-up
  Adolescent anxiety symptoms. The final score is represented by the T -score, that has a mean of 50 and a standard deviation of 10. With higher scores indicating more anxiety.
Working Alliance Inventory | Monthly during the six months of treatment.
  Quality of the therapeutic relationship. The WAI is scored on a 7-point Likert-type scale ranging from 1 (never) to 7 (always. Subscales can range from 12-83 and can be summed to obtain a total score-which range from 36-252. Higher scores reflect more positive ratings of the working alliance.
Service Utilization Questionnaire | Baseline
  Other services the youth may receive besides treatment conditions
Service Utilization Questionnaire | 3-month mid-treatment
  Other services the youth may receive besides treatment conditions
Service Utilization Questionnaire | 6-month end of treatment
  Other services the youth may receive besides treatment conditions
Service Utilization Questionnaire | 12-month follow-up
  Other services the youth may receive besides treatment conditions
Parent Adolescent Relationship Questionnaire (PARQ) | Baseline
  The PARQ is a psychometrically sound family functioning measure that is based on behavioral family systems therapy, and has been used in effectiveness research. Respondents are asked indicate if a statement that describes thoughts, feelings, and beliefs about their family is true or false. The PARQ items are summed to obtain a total score, with higher scores reflect more positive aspects of the parent-adolescent relationship.
Parent Adolescent Relationship Questionnaire (PARQ) | 6-month end of treatment
  The PARQ is a psychometrically sound family functioning measure that is based on behavioral family systems therapy, and has been used in effectiveness research. Respondents are asked indicate if a statement that describes thoughts, feelings, and beliefs about their family is true or false. The PARQ items are summed to obtain a total score, with higher scores reflect more positive aspects of the parent-adolescent relationship.
Parent Adolescent Relationship Questionnaire (PARQ) | 12-month follow-up
  The PARQ is a psychometrically sound family functioning measure that is based on behavioral family systems therapy, and has been used in effectiveness research. Respondents are asked indicate if a statement that describes thoughts, feelings, and beliefs about their family is true or false. The PARQ items are summed to obtain a total score, with higher scores reflect more positive aspects of the parent-adolescent relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Madisetti, Ph.D., Principal Investigator — Medical University of South Carolina; Phillippe B Cunningham, PhD, Principal Investigator — UTHealth
Locations (1):
- Division of Global and Community Health, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
At the expiration of the study locked data files and variable and scale dictionaries will be made available to the NIH for archiving and sharing with other researchers, in accordance with NIH policies. The Contact PI (Cunningham) will ensure that all datasets provided will be prepared in accordance with NHLBI requirements for data repository and associated documentation for submission to the Biological Specimen and Data Repository Information Coordinating Center; NHLBI Policy for Data Sharing from Clinical Trials and Epidemiological Studies; and NHLBI Guidelines for Data Set Preparation. Results from the proposed study will be presented in required reports to NIH. Additionally, results will be presented to clinical researchers, clinical treatment organizations, and state and national legislative bodies as requested. Within one year of completion of the study and publication of the main study findings we will make available the datasets publicly.

REFERENCES:
- [Background] Cunningham PB, Naar S, Roberts JR, Powell J, Ledgerwood DM, Randall J, Lozano BE, Halliday CA, Madisetti M, Ghosh S. Study protocol for clinical trial of the FIT Families multicomponent obesity intervention for African American adolescents and their caregivers: Next step from the ORBIT initiative. BMJ Open. 2024 Feb 13;14(2):e074552. doi: 10.1136/bmjopen-2023-074552. PMID 38355187
- [Background] Cunningham PB, Gilmore J, Naar S, Preston SD, Eubanks CF, Hubig NC, McClendon J, Ghosh S, Ryan-Pettes S. Opening the Black Box of Family-Based Treatments: An Artificial Intelligence Framework to Examine Therapeutic Alliance and Therapist Empathy. Clin Child Fam Psychol Rev. 2023 Dec;26(4):975-993. doi: 10.1007/s10567-023-00451-6. Epub 2023 Sep 7. PMID 37676364